CLINICAL TRIAL: NCT06139549
Title: The Effects of Playful Pathways, a Play-Based Developmentally Focused Group Program, and How it Affects Caregivers' Health Literacy and Self-Efficacy and Influences Outcomes for Infants
Brief Title: The Effects of Playful Pathways
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Arkansas Colleges of Health Education (Other)
Responsible Party: Principal Investigator, Allison Young, Assistant Professor, Arkansas Colleges of Health Education
Other Study IDs: ACHEFALL2023PP
Record Dates: First submitted 2023-09-17; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Gross Motor Development Delay
Keywords: INFANT; GROSS MOTOR DEVELOPMENT; GROUP SESSION

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Gross motor development group session — Group session for gross motor development

SUMMARY:
The purpose of this study is to evaluate infants ages 0-6 months of age before and after an 8 week developmental and educational "caregiver and baby" interactive program as well as 3 month following the conclusion of the program. The researchers aim to screen and identify developmental delays and the effects of the 8 week program on gross motor development as well as explore parent perceptions of the program.

The aim of this study is to assess the physical, social, and emotional outcomes of an interactive group program for infants 0-6 months and their families/caregiver.

ELIGIBILITY:
All babies typically developing or any diagnosis ages 0 - 6 months; parents/caregivers of babies typically developing or any diagnosis ages 0 - 6 months participating in the intervention. Sample size will be 12 babies ages 0-6 months and their caregivers (1-2 caregivers per baby). Total population 12 infants with up to 30 caregivers.

Inclusion criteria:

1. All babies typically developing or any diagnosis ages 0 - 6 months

Inclusion criteria for parents/caregivers:

1. At least 18 years of age
2. Able to communicate in and read English
3. Parent/caregiver of baby ages 0 - 6 months who is participating in the program
4. Ability to provide transportation to/from research site(s)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Infants ages 0-6 months Caregivers age 18 and older
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2023-11-08 (Estimated); Study Completion 2024-02-20 (Estimated)

PRIMARY OUTCOMES:
DAYC-2 | 9/20/23 - 2/20/24
  measure of gross motor development
PHLAT-8 | 9/20/23 - 2/20/24
  measure of health literacy

CONTACTS AND LOCATIONS:
Overall Officials: Allison N Young, DPT, Principal Investigator — Arkansas Colleges of Health Education
Locations (1):
- Arkansas Colleges of Health Education, Fort Smith, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alkhazrajy, L. A., & Aldeen, E. R. S. (2017). Assessment of mothers knowledge regarding the developmental milestone among children under two years in Iraq. American Journal of Applied Sciences, 14(9), 869-877.
- [Result] Aoyama T, Hikihara Y, Watanabe M, Wakabayashi H, Hanawa S, Omi N, Takimoto H, Tanaka S. Association Between Age of Achieving Gross Motor Development Milestones During Infancy and Body Fat Percentage at 6 to 7 Years of Age. Matern Child Health J. 2022 Feb;26(2):415-423. doi: 10.1007/s10995-021-03238-9. Epub 2021 Oct 16. PMID 34655425